CLINICAL TRIAL: NCT01433575
Title: A Single-center, Open-label, Single Dose, Randomized, Two-way Cross-over Study to Investigate the Pharmacokinetics, Safety, and Tolerability of RO4917838 in Healthy Chinese Volunteers
Brief Title: A Pharmacokinetic Study of RO4917838 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BP25274
Record Dates: First submitted 2011-08-31; First posted 2011-09-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (2):
- A (Experimental)
  Interventions: Drug: RO4917838
- B (Experimental)
  Interventions: Drug: RO4917838

INTERVENTIONS:
Drug: RO4917838 — 10 mg single oral dose
  Arms: A
Drug: RO4917838 — 20 mg single oral dose
  Arms: B

SUMMARY:
This single-center, open-label, single dose, randomized, two-way cross-over study will evaluate the pharmacokinetics, safety and tolerability of RO4917838 in healthy Chinese volunteers. Subjects will be randomized to receive a single oral dose of either 10 mg or 20 mg RO4917838 and, after a washout period of at least 21 but no more than 35 days, will be re-dosed with the alternative treatment. Anticipated time on study is up to 70 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male and female volunteers, 18 to 45 years of age inclusive at time of screening
* Healthy status is defined by absence of evidence of any active or chronic disease or disorder following a detailed medical and surgical history and a complete physical examination
* Body mass index (BMI) 19 to 28 kg/m2 inclusive

Exclusion Criteria:

* Pregnant or currently lactating females
* History of any clinically relevant disorder
* Any history of depressive episodes or treatment with antidepressants
* History of drug abuse within the past 2 years or positive results for drugs of abuse at screening or Day -1
* Alcohol dependence or history of this within the past 2 years or positive results for alcohol breath test at screening or Day -1
* Positive for HIV, hepatitis B or hepatitis C infection
* Regular smoker with consumption of more than 10 cigarettes a day or equivalent amount of tobacco
* Participation in a clinical study with an investigational drug or device within the last 3 months prior to dosing
* Medical history of significant drug allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | 12 days
Pharmacokinetics: Peak plasma concentrations (Cmax) | 12 days

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Beijing, China